CLINICAL TRIAL: NCT01190293
Title: A Pilot Evaluation of the Pharmacokinetics, Efficacy and Safety of Switching From Efavirenz to Maraviroc Administered at 600mg Then 300mg Twice-daily in Patients Suppressed on an Efavirenz-containing Regimen as Initial Therapy
Brief Title: PK Switch Efavirenz to Maraviroc in Patients Initially Suppressed on an Efavirenz-containing Regimen
Acronym: SSAT033
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 033
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All Subjects will receive the same intervention.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — All patients (previously on an efavirenz-based therapy) will be administered maraviroc at 600mg twice-daily for 2 weeks.
  Other Names: Efavirenz = Sustiva; Maraviroc = Celsentri

SUMMARY:
The purpose of the study aims is to help determine whether it is safe to change directly from efavirenz to maraviroc in patients who are stable on an efavirenz-containing regimen. The pharmacokinetics (drug levels) of efavirenz and maraviroc when efavirenz is stopped and maraviroc is started will be assessed.

Both the study patients and the study team will know which treatment is being taken at all times in the study.

DETAILED DESCRIPTION:
Maraviroc (MVC) is a CCR5 antagonist that prevents virus entry blocking the binding of R5-tropic HIV to the cell surface CCR5 co-receptor. The MERIT Study compared MVC with EFV, each with a Combivir backbone, as initial therapy. Using a non-inferiority margin of 10% MVC was non-inferior to EFV using the <400 copies/ml viral load cut-off but failed to reach non-inferiority when a <50 copies/ml analysis was used. Since this study was performed a more sensitive tropism assay has become routinely available and a re-analysis of the MERIT results showed that some of the patients with apparent R5-tropic virus actually had non-R5 virus. When these patients were excluded from the analysis, MVC did achieve non-inferiority compared to efavirenz. Of note, a subanalysis in the original MERIT Study of individuals with a baseline viral load below 100,000 copies/ml demonstrated only a small numerical difference between MVC and EFV recipients with 69.6% and 71.6% respectively achieving a viral load less than 50 copies/ml at 48 weeks. Recent data from the MOTIVATE Study (a comparison of maraviroc and placebo with optimised background regimen in treatment-experienced patients) showed geno2pheno (a genotypic algorithm for tropism estimation) to be as accurate as Trofile (a phenotypic assay) at predicting response to maraviroc. In situations where the genotypic and phenotypic test showed discordant results virological response was similar to where both demonstrated concordant R5-tropism.

Importantly MVC has been very well-tolerated in both treatment-naïve and treatment-experienced patients. Overall similar proportions of subjects experienced grade 3/4 adverse events; importantly, malignancy rates were similar in the two arms (4.4% on EFV and 2.8% on MVC). Broadly, individual adverse events occurred at similar frequencies in the two arms although abnormal dreams, dizziness and rash were all less common on MVC. In addition median lipid changes were greater in the EFV arm, correlating with a lower predicted risk of cardiovascular disease for MVC recipients.

Maraviroc is a substrate of the CYP3A4 enzyme; therefore, its metabolism is reduced by pure CYP3A4 inhibitors (most protease inhibitors) and increased by CYP3A4 inducers (such as EFV). Dose adjustments are required when MVC is co-administered with certain protease inhibitors (reduced from 300mg BD to 150mg BD) or EFV (increased from 300mg BD to 600mg BD). When switching from a protease inhibitor (PI), the PI is cleared rapidly such that no interim dose adjustment would be required. EFV, however, is cleared slowly and can remain at detectable concentrations for several days and can continue to induce CYP3A4 for some time after stopping the drug. Therefore, if switching from EFV to MVC, it can be expected that EFV may affect MVC concentrations for a period of time after the switch. The length of time that the inducing effect of EFV will persist for after stopping the drug is unclear. Crucially, the inducing effect of EFV could result in sub-therapeutic MVC concentrations (if MVC is started immediately after efavirenz) during initial therapy. Sub-therapeutic drug concentrations are associated with virological failure and development of resistance. In addition, maintaining an elevated dose of MVC after the induction effect of EFV has worn off could result in adverse events (such as hypotension) hence the fact that, in this study, increased dose will be maintained for a 2 week period only.

In conclusion, while MVC dose adjustments required during co-administration with EFV are clear, the correct dose of MVC when switching from an EFV-containing regimen remains unknown.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 56 days prior to the baseline visit:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedure and must be willing to comply with all study requirements.
2. Males or non-pregnant, non-lactating females.
3. Between 18 to 65 years, inclusive.
4. Documented HIV-1 infection of at least 6 months duration.
5. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study.
6. CD4 count > 50 cells/mm3 at screening (Note retesting of screening CD4 count is allowed).
7. Receiving an antiretroviral regimen including two NRTI with efavirenz, without any history of virological failure and agrees to remain on this regimen unless change is clinically indicated (history of drug switches is allowed only if the reason was tolerability/toxicity/convenience of dosing).
8. Viral load <50 copies/ml at screening and for at least 12 weeks prior to screening visit (Note retesting of screening viral load is allowed).
9. R5-tropic virus as determined by genotypic assay performed at screening visit.
10. No medical, psychiatric or substance misuse disorders felt by the investigator to impact on the subject's ability to participate in the study including a positive drugs of abuse test. (Note: a positive test for cannabinoids will not exclude the subject from the study).

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Dual, mixed or X4-tropic virus on geno2pheno tropism sample
2. HIV-2 co-infection
3. Any prior CCR5 antagonists
4. Any genotypic resistance to NNRTI or backbone NRTI on screening or prior tests (or likely from treatment history)
5. Disallowed concomitant medication as per the SPC for Celsentri or components of NRTI backbone (see section 5.1.1)
6. Any medical condition or psychiatric illness that may, in the opinion of the investigator, affect patient safety or the integrity of the results
7. ALT or AST elevation greater than five times the upper limit of normal
8. Estimated GFR (MDRD) less than 50ml/min
9. Hepatitis B or C co-infection (defined as positive hepatitis B surface antigen or detectable hepatitis C RNA; hepatitis C antibody positive individuals with undetectable RNA will be eligible for inclusion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pharmocokinetics of maraviroc dosed at 600mg followed by 300mg thereafter following cessation of efavirenz 600mg. | 2 weeks
  To assess the pharmacokinetics of maraviroc administered at 600mg twice-daily for 2 weeks to male and female HIV-1 infected patients who have achieved viral suppression on efavirenz-based therapy followed by maraviroc 300mg twice-daily until the end of the study.

SECONDARY OUTCOMES:
Virological suppression and CD4 rise | 4 weeks
  To assess the maintenance of virological suppression and CD4 rise when switching efavirenz to maraviroc.
Safety and tolerability of an efavirenz to maraviroc switch. | 24 weeks
  To assess the safety and tolerability of switching from efavirenz to maraviroc.
Genetic influence | 24 weeks
  To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Waters, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom

REFERENCES:
- See also: (St Stephen's AIDS Trust website) — http://www.ssat.org.uk/